CLINICAL TRIAL: NCT04352569
Title: Efficacy of tDCS in the Treatment of Resistant Auditory Hallucinations in Schizophrenia: A Double Blind, Randomized Controlled Study
Brief Title: Efficacy of tDCS in the Treatment of Resistant Auditory Hallucinations in Schizophrenia
Acronym: TDCSHALLU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de Ville-Evrard, France (Other)
Responsible Party: Principal Investigator, Noomane Bouaziz, MD, MD, Centre hospitalier de Ville-Evrard, France
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DMDPT-TCH/MM/2015-A00842-47
Record Dates: First submitted 2015-10-27; First posted 2020-04-20 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Schizophrenia; Hallucinations; Refractory Schizophrenia
MeSH Terms: conditions — Schizophrenia; Hallucinations; Schizophrenia, Treatment-Resistant | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- transcranial direct current stimulation (Active Comparator): The transcranial direct current stimulation (tDCS) with two elecrodes placed over the scalp: the anode over the LTP, le cathode over L DLPFG.
  Interventions: Device: transcranial direct current stimulation
- transcranial direct current stimulation sham (Sham Comparator): tDCS device allows sham stimulation. This technic give the same impression that active stimulation and allows optimum placebo stimulation.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — transcranial direct current stimulation (tDCS) is a non invasive brain stimulation technic
  Other Names: tDCS

SUMMARY:
The regions which are assumed to underlie the pathophysiology of schizophrenia, namely hypoactivity at the prefrontal level and pathological hyperactivity of the associative regions of the language located in the left temporoparietal region.

To assess the efficacy of tDCS on auditory hallucinations, the investigators performs an randomized double blind versus placebo trial. In each arms patients will receive two tDCS sessions a day during two weeks.

DETAILED DESCRIPTION:
Hearing hallucinations are one of the major symptoms of schizophrenia. In 30% of patients they are resistant to common psychotropic treatments. tDCS (Transcranial Direct Current Stimulation) is a technical of brain stimulation, non-invasive, painless that modulates brain activity by the transcranial administration of a low-intensity electric current, via two electrodes (an anode and a cathode). Several scientifics studies have reported a beneficial effect of tDCS in the treatment of pain, depression and especially hearing hallucinations in schizophrenia.

The main study purpose is to evaluate the effectiveness of tDCS on resistant auditory hallucinations in patients with schizophrenia.

Then, to evaluate the effectiveness of tDCS on global schizophrenic symptomatology and to assess the impact of tDCS on patients' quality of life.

Also the study, evaluate the impact of tDCS on cortical excitability. We measure the change in serum BDNF (Brain Derived Neutrophic Factor) before and after tDCS stimulation. Indeed, to evaluate the impact of tDCS on neurocognitive functions.

Patients will receive either active tDCS or placebo tDCS randomly. All patients will have two tDCS/day sessions, one hour apart, for 2 working weeks. The stimulation parameters will be consistent with the literature data, namely: Intensity = 2mA; duration of sessions = 20 minutes; total number of sessions = 20 (2 daily sessions for two working weeks).

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia according to DSM-V.
* Refractory auditory hallucinations(despite two antipsychotics trials).
* Right-handed patients.
* Written informed consent.

Exclusion Criteria:

* Presence of other psychiatric disorders than schizophrenia (except addiction to tobacco or caffeine ).
* History of severe head trauma or coma.
* History of epilepsy or neurological disorder or a general medical condition.
* Presence of intracranial metallic objects or pacemaker.
* Hospitalized patients without consent.
* pregnant women .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2016-05-03 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
auditory hallucinations rating scale (AHRS) | At baseline
  AHRS is a scale frequently used to assess auditory hallucinations in schizophrenia studies (Hoffman et al. 2005).
auditory hallucinations rating scale (AHRS) | 15 days after
  AHRS is a scale frequently used to assess auditory hallucinations in schizophrenia studies (Hoffman et al. 2005).

SECONDARY OUTCOMES:
PANSS, | At baseline
  Positive and negative symptom scale (PANSS, Kay et al. 1988)
PANSS, | 15 days after
  Positive and negative symptom scale (PANSS, Kay et al. 1988)
CGI | At baseline
  clinical global impression (Kadouri et al. 2007)
CGI | 15 days after
  clinical global impression (Kadouri et al. 2007)

CONTACTS AND LOCATIONS:
Overall Officials: NOOMANE BOUAZIZ, MD, Principal Investigator — Unité de Recherche Clinique de l'EPS de Ville Evard
Locations (1):
- unité de recherche clinique de l'E.P.S de Ville Evrard, Neuilly-sur-Marne, France

IPD SHARING:
Plan to Share IPD: Undecided